CLINICAL TRIAL: NCT02392169
Title: Relationship Between the Neuroendocrine Substrates, Candidate Genes and Endophenotypes in Patients With Attention-deficit/Hyperactivity Disorder
Brief Title: Neuroendocrine Substrates, Candidate Genes and Endophenotypes in ADHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Liang-Jen, Associate Professor and Visiting Staff, Chang Gung Memorial Hospital
Other Study IDs: 101-4835A3
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: neuroendocrine; ADHD; heredity; cognitive function
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — oral mucosal cells
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Methylphenidate — Patients used Retina or Concerta twice a day lasting for one year.
  Other Names: Retalin, concerta

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is one of the most common child and adolescent psychiatric disorders. In recent years, some researchers have become interested in analyzing neuroendocrine substrate levels in ADHD, including dehydroepiandrosterone (DHEA), dehydroepiandrosterone sulfate (DHEA-S), cortisol and testosterone. Previous work in ADHD has established a strong heritable component to the phenotype. The STS gene, SULT2A1 gene and TH gene are associated with the function of DHEA/DHEA-S, and the NR3C1 gene is associated with the regulation of cortisol. Therefore, the relationship between these genes and the etiology of ADHD warrants investigation. Moreover, compared to the phenotype, the endophenotypes of ADHD may be more capable of detecting the underlying neurobiological and hereditary mechanisms. Therefore, this study aims to investigate the relationships between neuroendocrine substrates (DHEA, DHEA-S, cortisol and testosterone), candidate genes (STS gene, SULT2A1 gene, TH gene and NR3C1 gene) and the phenotype and endophenotypes (disease subtypes, neurocognitive function and response to treatment) of ADHD.

To complete this work, we will recruit 300 patients with ADHD (probands) and 600 biological parents of the probands. DNA will be extracted from buccal cells by cheek swab. At baseline, saliva samples of ADHD patients will be collected between 7:00 and 8:00 am using the passive drool method, to analyze the levels of neuroendocrine substrates. The patients will undergo assessment for their clinical symptoms and neurocognitive function. Methylphenidate will then be administered to the patients and the usual practice followed. At week 4 and week 52, procedures similar to those performed at baseline will be repeated.

The results of this study may further elucidate the complexity of the pathophysiology of ADHD. We may determine whether the neuroendocrine system, which contains levels of neuroendocrine substrates and associated genes, plays a crucial role in the phenotype and endophenotypes of ADHD. The information may serve as an important reference for the direction of future study and clinical treatment for patients with ADHD.

DETAILED DESCRIPTION:
1. We will recruit the patients who meet the criteria for ADHD outlined in the DSM-IV. The diagnosis will be made by a child psychiatrist in a structured interview using the Kiddie Epidemiologic Version of the Schedule for Affective Disorders and Schizophrenia (K-SADS-E ).
2. The variables of questionnaire from interview include the personal data as below: Age, gender, family background, the significant pressure on growth, positions and incomes of parents, and the process of mother's pregnant.
3. For genotyping analysis, DNA of patients and their biological parents will be collected using cheek swab to collect oral mucosal cells, then put it in the refrigerator at-80°C. The genotyping of STS gene, SULT2A1 gene, TH gene and NR3C1 gene will be identified.
4. The saliva of patients with ADHD will be collected by passive drool method at 7:00-8:00 in the morning. The saliva specimen which use to analysis endocrine substance concentration should be placed at - 80 ° C freezer as soon as possible.
5. The psychiatrist or psychologist will rate patients' symptom severity of the case. The parents of the patients have to fill in the ASRS, SNAP-IV(parent form) and CBCL. The teacher of the case has to fill in the SNAP-IV(teacher form) and TRF. The patients were administered the computerized CPT in a room dedicated to the testing to minimize the variability of the test conditions.
6. After the initial assessment, patients with ADHD will begin to receive methylphenidate (MPH) treatment. Patient care was left to the discretion of the psychiatrists, who were given no treatment instructions and simply encouraged to manage their patients according to usual practice. Dosage and drug form can be adjust through the height and weight of the case and his/her clinical needs. The times and frequency of track back should be reference the clinical needs, patients and their parents' willingness. During the follow-up, non-drug therapy. (e.g. Behavioral therapy, Sensory integration therapy) will not be restricted. If the patients whose condition needs to be treated with drugs other than MPH, the tests must be discontinued.
7. After four weeks, we will assess the short-term efficacy symptoms and cognitive function of the patients. Patients will be saked to collect saliva at 7:00-8:00 in the morning¸ after that, to analysis endocrine substance concentration. The behavioral and neurocognitive assessment will be performed using CGI-S、SNAP-IV(parent form), SNAP-IV(teacher form), CBCL, TRF and CPT.
8. At week 52, we will assess the long-term efficacy of the cases the symptoms and cognitive function in the first 52 weeks. We will collect the saliva sampe of ADHD patients at 7:00-8:00 in the morning. The behavioral and neurocognitive assessment will be performed using CGI-S、SNAP-IV(parent form), SNAP-IV(teacher form), CBCL, TRF, CPT and WISC-IV.

   Finally, in K-SADS-E interviews to assess whether the patient is still meet the ADHD diagnostic criteria of DSM-IV-TR.
9. Saliva sample will be collected into collecting tubes and stored in the refrigerator at-80°C. The salivary levels of DHEA, DHREA-S, cortisol and testosterone will be determined using ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADHD aged between 6 and 16.
* The patients were either newly diagnosed with ADHD or had an existing diagnosis but had not taken medication for ADHD during the previous 6 months or more.

Exclusion Criteria:

* Patients with a history of major physical or additional psychiatric diseases .

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients from Kaohsiung, Taiwan by specialist clinical diagnosis of ADHD.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The Chinese version of Swanson, Nolan and Pelham IV Scale (SNAP-IV) | 15 min

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Jen Wang, MD, MPH, Principal Investigator — Chang Gung Memorial Hospital, Kaohsiung, Taiwan
Locations (1):
- Liang-Jen Wang, Kaohsiung City, Kaohsiung, Taiwan